CLINICAL TRIAL: NCT05973071
Title: Clinical Use of a Contraceptive Decision Aid and Patient Outcomes: An Experimental Clinical Trial
Brief Title: Clinical Use of a Contraceptive Decision Aid and Patient Outcomes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas Christian University (Other)
Collaborators: Oklahoma State University (Other)
Responsible Party: Principal Investigator, Sarah Hill, Professor, Texas Christian University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TCU020519782
Record Dates: First submitted 2023-06-15; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Contraceptive Usage
Keywords: Decision Aid
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be block assigned to either the Tuune condition or the traditional contraceptive counseling condition.
Who Masked: Outcomes Assessor
Masking Description: All data will be analyzed by a blind coding process, meaning that the researcher performing the analyses will be unaware of our research hypotheses. All date and timestamp information will also be removed to ensure that those analyzing the data cannot infer which patients were in the Tuune condition and which received a traditional patient appointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tuune (Experimental): Participants complete the Tuune contraceptive decision aid health questionnaire as part of their standard OBGYN clinic appointment.
  Interventions: Behavioral: Tuune Supplemented Contraceptive Visit
- Control (Active Comparator): Participants will complete a standard OBGYN clinic appointment without using the Tuune contraceptive decision aid health questionnaire.
  Interventions: Behavioral: Traditional Contraceptive Visit

INTERVENTIONS:
Behavioral: Tuune Supplemented Contraceptive Visit — Participants complete the Tuune contraceptive decision aid health questionnaire (Tuune for clinics) as part of their standard OBGYN clinic appointment.
  Arms: Tuune
Behavioral: Traditional Contraceptive Visit — Participants will complete a standard OBGYN clinic appointment without using the Tuune contraceptive decision aid health questionnaire (Tuune for Clinics).
  Arms: Control

SUMMARY:
The study at hand aims to examine whether incorporating use of a contraceptive decision aid (Tuune for Clinics) improves outcomes for patients seeking contraceptive care. To achieve this the investigators will test: the hypothesis that use of the Tuune decision aid in contraceptive care appointments will: (a) improve patient satisfaction, (b) increase patient positivity toward contraceptive use, and (c) improve patient outcomes, including: (ci) greater adherence to their prescribed contraceptive and (cii) fewer negative side-effects, relative to that which is observed for patients receiving a contraceptive recommendation from a traditional contraceptive counseling appointment.

DETAILED DESCRIPTION:
Participants: Participants will be block assigned to one of two groups, an experimental and a control group. In the experimental group, women will discuss the Tuune contraception recommendations with their physician during their contraceptive counseling appointment. In the control group, women will go through a traditional counseling appointment with their physician.

Materials and Procedure: Participants will be block-randomized to either the traditional contraceptive counseling appointment or to the Tuune facilitated contraceptive counseling appointment. Data for the control condition will be collected prior to data collection for the Tuune condition to avoid introducing bias or contaminating the control condition viz care provider increase in contraceptive knowledge as a result of using Tuune. Once 200 patients have been successfully recruited and processed in the control condition, the clinic will incorporate use of the Tuune decision aid into patient appointments until such a time that 200 patients are successfully recruited and processed. Patients scheduling appointments with OSU Obstetrics and Gynecology during the intervention period (i.e., during the period in which use of the Tuune decision aid is being incorporated into patient appointments) will be sent a QR code in advance of their appointment that allows them to access the Tuune decision aid. Participants will be instructed to complete the decision aid health questionnaire (which asks patients to report on health conditions, as in a typical patient intake form, in addition to numerous questions about hormonal conditions and contraception goals) in advance of their appointment. Participants in the control condition will simply be asked standard clinic intake questions per a typical patient appointment.

All participants will be recruited by clinic staff at the time of their appointment. Prospective participants will be informed that they must be between the ages of 18 and 50 years old and cannot be pregnant, breastfeeding, or wishing to become pregnant. All participants will read over the recruitment materials and consent form in the waiting room of the clinic when waiting for their appointment. The nurse attending to patients will then go over the consent form to answer any questions for participants wishing to participate. All participants will then meet with their contraceptive care provider and discuss their reproductive health and contraceptive options. In the traditional appointment group, physicians will proceed as they normally would. In the Tuune condition, physicians will discuss the results of the Tuune health assessment with their patients by going through all the hormonal contraceptive suggestions provided by the digital aide, answering any questions, and providing additional information and guidance per the patient's needs.

Both groups of participants will be given a QR code that will take them to a brief survey to assess their satisfaction with their care, the degree to which they perceived their care to be person-centered, their positivity toward the medication they had been prescribed, and their perceived likelihood that they will take the prescribed medication. Finally, participants will be asked for their contact information for follow-up purposes and for delivery of a $10 digital gift card that will be sent to participants' phone or email as a thank you for their participation.

Three months after the contraceptive counseling appointment, participants will be contacted via email or text using the contact information provided at the time of their patient appointment to complete a brief follow-up survey in exchange for a $15 digital gift card. Three months was chosen as the follow-up period because it takes about three months for the body to adjust to a new hormonal contraceptive and for initial side effects to subside. Participants will be asked about whether they are still on the prescribed contraceptive and about their adherence and positivity toward the prescribed contraceptive. Participants will also be asked to report the number of side effects that improved and the number of side effects that worsened since beginning the recommended contraception.

The exact items and scoring procedures for all measures to be used can be viewed on the Open Science Framework (Open Science Project Number: 3hdm6). In particular, at Time 1 (immediately following the patient appointment) the investigators will assess: (a) patient satisfaction, (b) perceptions of the degree to which they received person-centered contraceptive counseling (PCCC), (c) positivity toward their prescribed medication, and (d) contraceptive use expectations. At Time 2 (3 months post-appointment), the investigators will assess (e) whether patients are still using their prescribed contraception, (f) their adherence to their contraception medication, and (g) their experience with both positive and negative side effects. Each of the chosen scales has been shown to be reliable and valid in a variety of clinical and non-clinical settings. Minor modifications to some established scales were made for the purposes of making them tailored to research question at hand (see Open Science Project Number 3hdm6 for details).

All materials and methods for this project are pre-registered and available on the Open Science Framework (Project: 3hdm6 available here: https://osf.io/3hdm6/).

Data Handling: All data will be analyzed by a blind coding process, meaning that the researchers performing the data analyses and the PI will be blind to which condition participants are in prior to data analysis. To this end all date and timestamp information will be removed by a trained scientist who is not affiliated with the current project and who is blind to the nature of the hypothesis under investigation. This will help ensure that those analyzing the data cannot infer which patients were in the Tuune condition and which received a traditional patient appointment.

Expected Outcomes: The investigators expect that patients using the Tuune decision aid will exhibit higher levels of patient satisfaction and greater positivity toward their prescribed contraceptive than women who receive a traditional contraceptive appointment only. Further, the investigators expect that patients using the Tuune decision aid will exhibit higher rates of contraceptive continuity, greater adherence to their prescription, and will report fewer negative side effects than those in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* New or existing patients at Oklahoma State University OBGYN seeking contraceptive counseling.
* Native Speakers of English.

Exclusion Criteria:

* Women who are currently pregnant or breastfeeding
* Women who wish to become pregnant within the next 12 months

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction & Appointment Evaluation [1] | Administered at immediate follow-up.
  This scale measures patient satisfaction with a contraceptive counseling appointment. Items include "Overall, I was satisfied with the birth control counselling," and "The session helped to strengthen my confidence in my method of birth control." Scale values range from 1 = Strongly agree to 7 = Strongly disagree. Item 10 needs to be reverse coded (R). An overall score can be created for this measure by averaging items.
  All items could not be pasted in this description box due to character limit. The full list of items is available at https://osf.io/3hdm6/.
Patient Satisfaction [2] | Administered at immediate follow-up.
  This single item measures patient satisfaction with the birth control services received from healthcare providers.
  Scoring Instructions: Scale values range from 1 = Not at all satisfied to 7 = Extremely satisfied.
  1. In general, how satisfied or dissatisfied would you say you are with the birth control services you have received from healthcare providers?
Person Centered Contraceptive Counseling (PCCC) [3] | Administered at immediate follow-up.
  This measure is an evaluation of whether the physician provided person-centered contraceptive counseling.
  Scoring Instructions: An overall score can be created for this measure by averaging items. Scale values range from 1 = Poor to 4 = Very good. No items need to be reverse coded.
  Think about your visit. How do you think [provider name] did? Please rate them on each of the following by circling a number (1 = Poor, 2 = Fair, 3 = Good, 4 = Very good).
  1. Respecting me as a person.
  2. Letting me say what mattered to me about my birth control method.
  3. Taking my preferences about my birth control seriously.
  4. Giving me enough information to make the best decision about my birth control method.
Positivity Toward Their Prescribed Medication [4] | Administered at immediate follow-up
  This scale measures patient positivity toward the prescribed medication.
  Scoring Instructions: An overall score can be created for this measure by averaging items. Scale values range from 1 = Not at all to 7 = Extremely. Item 2 needs to be reverse coded (R).
  1. How positively do you feel about this medication?
  2. How negatively do you feel about this medication? (R)
Contraceptive Use Expectations [4] | Administered at immediate follow-up
  This scale measures the patient's perceived likelihood that they will take the prescribed medication.
  Scoring Instructions: Scale values range from 1 = Not at all to 7 = Extremely.
  1.How likely are you to take this medication?

SECONDARY OUTCOMES:
Post-Appointment Contraceptive Adherence [5,6] | Administered at 3 month digital follow-up
  This scale measures participants' degree of adherence to the prescribed medication since beginning their recommended birth control. Some example items are "Do you sometimes forget to take your birth control?" and "How often do you have difficulty remembering to take your birth control?" Items 1 - 7 have a yes/no response format (No = 1, Yes = 0). Item 5 needs to be reverse coded (R). Scale values for item 8 range from 0 = Never/Rarely to 4 = All the time. To standardized item 8, we will divide the result by 4. All items will be summed to create a continuous measure of self-reported adherence ranging from 0 - 8 with higher values corresponding to higher adherence.
  All items could not be pasted in this description box due to character limit. The full list of items is available at https://osf.io/3hdm6/.
Positivity Toward Their Prescribed Medication [4] | Administered at 3 month digital follow-up
  This scale measures patient positivity toward the prescribed medication.
  Scoring Instructions: An overall score can be created for this measure by averaging items. Scale values range from 1 = Not at all to 7 = Extremely. Item 2 needs to be reverse coded (R).
  1. How positively do you feel about this medication?
  2. How negatively do you feel about this medication? (R)
Patient Experiences with their Birth Control | Administered at 3 month digital follow-up.
  These items ask about patient experiences on their birth control.
  Scoring Instructions: The following items will be loaded into a Multivariate Analysis of Variance (MANOVA). Scale values range from 1 = Strongly agree to 7 = Strongly disagree. Item 1 needs to be reverse coded (R).
  1. I have experienced unpleasant side effects from my birth control. (R)
  2. I feel better on my birth control than I felt when off of it.
  3. I am happy with the birth control option I chose.
  4. I plan to continue using my current birth control.
Patient Experiences with their Birth Control - Side Effects | Administered at 3 month digital follow-up.
  Participants will be presented with a list of side effects (available at https://osf.io/3hdm6/) and asked to select which have improved/worsened since starting the recommended birth control. These items will be summed to determine 1) the number of side effects that improved since the participant began the recommended birth control and 2) the number of side effects that worsened since the participant began the recommended birth control.
  Scoring Instructions: To calculate a score for each item sum the number of side effects indicated by the respondent.
  Below is a list of side effects often associated with birth control. Since starting your birth control…
  1. Which of the following side effects have improved? [Select all that apply]
  2. Which of the following side effects have worsened? [Select all that apply]
Post Appointment Contraceptive Use | Administered at 3 month digital follow-up.
  This items measures participant discontinuation rate from their prescribed method of birth control.
  Scoring Instructions: This item has a yes/no response format.
  1. I am still using the birth control I was prescribed at my appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah E Hill, PhD, Principal Investigator — Texas Christian University
Locations (1):
- Texas Christian University, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bitzer J, Oppelt PG, Deten A. Evaluation of a patient-centred, needs-based approach to support shared decision making in contraceptive counselling: the COCO study. Eur J Contracept Reprod Health Care. 2021 Aug;26(4):326-333. doi: 10.1080/13625187.2021.1908539. Epub 2021 Apr 19. PMID 33871288
- [Background] Oakley LP, Harvey SM, Lopez-Cevallos DF. Racial and Ethnic Discrimination, Medical Mistrust, and Satisfaction with Birth Control Services among Young Adult Latinas. Womens Health Issues. 2018 Jul-Aug;28(4):313-320. doi: 10.1016/j.whi.2018.03.007. Epub 2018 May 2. PMID 29729838
- [Background] Dehlendorf C, Fox E, Silverstein IA, Hoffman A, Campora Perez MP, Holt K, Reed R, Hessler D. Development of the Person-Centered Contraceptive Counseling scale (PCCC), a short form of the Interpersonal Quality of Family Planning care scale. Contraception. 2021 May;103(5):310-315. doi: 10.1016/j.contraception.2021.01.008. Epub 2021 Jan 27. PMID 33508252
- [Background] Minton AR, Young NA, Nievera MA, Mikels JA. Positivity helps the medicine go down: Leveraging framing and affective contexts to enhance the likelihood to take medications. Emotion. 2021 Aug;21(5):1062-1073. doi: 10.1037/emo0000798. Epub 2020 Nov 12. PMID 33180530
- [Background] Morisky DE, Ang A, Krousel-Wood M, Ward HJ. Predictive validity of a medication adherence measure in an outpatient setting. J Clin Hypertens (Greenwich). 2008 May;10(5):348-54. doi: 10.1111/j.1751-7176.2008.07572.x. PMID 18453793
- [Background] Tomaszewski D, Aronson BD, Kading M, Morisky D. Relationship between self-efficacy and patient knowledge on adherence to oral contraceptives using the Morisky Medication Adherence Scale (MMAS-8). Reprod Health. 2017 Sep 6;14(1):110. doi: 10.1186/s12978-017-0374-6. PMID 28874178